CLINICAL TRIAL: NCT05558891
Title: THRIVE: Pilot Study of a Brief, Recovery-focused Intervention for Crisis Stabilization Centers
Brief Title: Pilot Study of a Brief, Recovery-focused Intervention for Crisis Stabilization Centers
Acronym: THRIVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centerstone Research Institute (Other)
Collaborators: University of Rochester (Other)
Responsible Party: Principal Investigator, Jordan Nelon, Director of Evaluation Science, Centerstone Research Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CenterstoneRI; YIG-0-113-20 (Other Grant/Funding Number: American Foundation for Suicide Prevention)
Record Dates: First submitted 2022-06-30; First posted 2022-09-28 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Suicide
MeSH Terms: conditions — Suicide | interventions — Nicotine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: THRIVE + Usual Care (Experimental): Individuals presenting to a community-based crisis stabilization center who are age 18-plus and screen positive for suicide risk
  Interventions: Behavioral: THRIVE; Behavioral: Usual Care
- Usual Care (Active Comparator): Individuals presenting to a community-based crisis stabilization center who are age 18-plus and screen positive for suicide risk
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: THRIVE — Toward Hope, Recovery, Interpersonal Relationships, Values and Engagement (THRIVE), is a brief, suicide-specific, narrative, recovery-focused, 60 minute intervention. THRIVE includes three components: 1) Sharing the suicide narrative; 2) Completing the Lifeline and Meaning Reconstruction; 3) Completing the Meaningful Living Plan (MLP).
  Arms: Experimental: THRIVE + Usual Care
Behavioral: Usual Care — Care as Usual in this Crisis Stabilization Unit includes medication management, medication management, safety planning Intervention, group psychoeducation, discharge planning, and community linkages

SUMMARY:
Crisis Stabilization Centers (CSCs) have a unique role to play in Emergency Department diversion and suicide-specific care. However, brief interventions tailored for CSC settings are needed. This study will examine a new, 60-minute, narrative, technology-based, recovery-oriented intervention called THRIVE. THRIVE may help people make meaning of their suicide crisis, reduce suicidal ideation, and increase their recovery compared to usual care. If effective, THRIVE will help CSCs deliver better recovery-focused care.

DETAILED DESCRIPTION:
More than 5.3 million individuals at risk for suicide seek treatment through emergency departments (EDs) each year despite the fact that EDs are not well suited for their care. Crisis Stabilization Centers (CSCs) have been proposed as a person-centered alternative to EDs. More than 600 CSCs nationwide operate 24 hours per day, accept walk-ins, provide care regardless of ability to pay, and partner with local law enforcement to divert suicidal patients from EDs. However, research outcomes on CSCs are mixed, likely associated with the fact that brief, recovery-oriented interventions with the potency to decrease suicide attempts and deaths are needed in CSCs but do not exist. Toward recovery, hope, recovery, interpersonal growth, values, and engagement (THRIVE) is a 60 minute intervention developed by the Principal Investigator and CSC stakeholders. THRIVE is uniquely tailored to CSC workflows and helps guests increase hopefulness, make meaning from stressful life events, and promote self-efficacy to prevent suicide attempts. In THRIVE, the guest is asked to narrate the suicide crisis, make meaning of the crisis through building an autobiographical timeline, and construct actionable future goals through an building an interactive meaningful living plan. THRIVE is conducted via a tablet so that all materials can be saved electronically in a HIPAA-compliant cloud to support providers in collaborating on care goals during and after discharge. The goal of this project is to fill a critical gap in the crisis stabilization literature by testing THRIVE as a novel solution to maximize the effectiveness of CSCs. This study will address the following aims: 1) Examine the feasibility, acceptability, and ecological validity of THRIVE as a unique fit for CSC guests (n = 30) and staff; 2) Conduct a pilot randomized trial (n = 150) to examine the degree to which THRIVE engages proposed recovery-oriented mechanisms of change relevant to the unique treatment philosophies of CSC settings; 3) As part of the pilot randomized trial, compare the outcomes of THRIVE + Usual Care (THRIVE + UC) to the outcomes of Usual Care (UC) delivered in the CSC (i.e., on recovery orientation, suicidal ideation, resolved suicide plans and preparation, treatment engagement, and acute psychiatric re-admissions). In Phase I (Aim 1), participants will be administered quantitative surveys after experiencing the THRIVE intervention. In Phase II (Aims, 2-3), participants in the RCT will be administered surveys at baseline, discharge, 1 month follow-up, and 3-month follow-up time points. CSCs represent the future of suicide-specific care and THRIVE is a novel intervention with the potential to impact more than 5.3 million individuals in a highly lethal group - suicidal individuals seeking care at EDs diverted to CSCs.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to the crisis stabilization center (CSC)
* Davidson county resident
* English-speaking
* Able to provide informed consent
* Willing to complete a locator form for follow-up assessments
* Willing to complete two emergency contacts
* Medically and clinically cleared by onsite psychiatrist/nurse practitioner
* Increased risk for suicide (Patient safety screener-3, Item 2 and/or 3 is "Yes")
* Willing and able to discuss their experiences around suicidal thoughts and/or attempts

Exclusion Criteria:

* Individuals who are acutely psychotic
* Individuals unable to communicate with the research team

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2022-06-22 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Meaning made of stress | 3 months
  Integration of Stressful Life Experiences Scale (ISLES; Holland et al., 2010). Subscale scores range from 11 to 55 (Footing in the World subscale), 5 to 25 (Comprehensibility subscale) and 16 to 80 (Total ISLES score). Higher scores on each ISLES subscale and the ISLES total score represent greater meaning reconstruction.
Hopefulness | 3 months
  Adult State Hope Scale (ASHS; Snyder et al., 1996). Subscale scores range from 3 to 34 (Pathways subscale), from 3 to 24 (Agency subscale), and from 6 to 48 (Total Hope Score). Higher scores on each ASHS subscale and the ASHS total score represent higher levels of hope.
Self-efficacy to avoid suicidal action | 3 months
  Self-Efficacy to Avoid Suicidal Action Scale (SEASA; Czyz et al., 2014). The total score on the SEASA ranges from 0 to 54, with higher levels presenting higher self-efficacy to avoid suicidal action.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Lockman, PhD, Principal Investigator — Centerstone Research Institute
Locations (1):
- Mental Health Cooperative, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lockman JD, Pisani AR, Angerer BP, Graham AC, Henry J, Lloyd F. THRIVE: Feasibility, Acceptability, and Social Validity of a Brief Recovery-Focused Intervention in Crisis Stabilization Centers. Suicide Life Threat Behav. 2025 Jun;55(3):e70021. doi: 10.1111/sltb.70021. PMID 40401321